CLINICAL TRIAL: NCT02221193
Title: Site-Specific Mouth Rinsing to Improve Oral Odor by Altering Bacterial Counts: Blind Crossover Clinical Study
Brief Title: Comparing Site Specific Mouth Disinfection With Commercial Oral Mouth Rinse With Traditional Oral Maouth Disinfection
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Al-Baha University (Other)
Responsible Party: Principal Investigator, Dr Mohammed Abdullah Alqumber, Assistant Professor, Al-Baha University
Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0568677142
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Oral Odor (Halitosis); The Study Want to Know if Site Specific Mouth Rinsing With Oral Mouth Disinfectants Can be Better Than Paonoral Mouth Rinsing
MeSH Terms: conditions — Halitosis | interventions — Crossing Over, Genetic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- site specific vs panoral disinfection (Experimental)
  Interventions: Other: traditional mouth rinsing and site-specific mouth rinsing (crossover)

INTERVENTIONS:
Other: traditional mouth rinsing and site-specific mouth rinsing (crossover) — blinded prospective, descriptive correlational crossover cross-section clinical trial conduct during the month of Ramadan in the lunar Hajri year 1434 AH (10 July 2013-8 August 2013) in Albaha province in Saudi Arabia involving the application of Listerine® Cool Mint® mouth rinse by either the traditional panoral rinsing method or a site-specific disinfection method targeting the subgingival and supragingival plaque and the posterior third of the tongue dorsum while avoiding the remaining locations within the oral cavity

SUMMARY:
Objectives: To determine whether site-specific mouth rinsing with oral disinfectants can improve oral odor beyond the traditional panoral mouth disinfection with mouth rinses by targeting specifically oral malodor implicate anaerobic bacteria.

Methods: Twenty healthy fasting subjects volunteered for a blinded prospective, descriptive correlational crossover cross-section clinical trial conduct during the month of Ramadan in the lunar Hajri year 1434 AH (10 July 2013-8 August 2013) in Albaha province in Saudi Arabia involving the application of Listerine® Cool Mint® mouth rinse by either the traditional panoral rinsing method or a site-specific disinfection method targeting the subgingival and supragingival plaque and the posterior third of the tongue dorsum while avoiding the remaining locations within the oral cavity. The viable anaerobic and aerobic bacterial counts, volatile sulfur compounds (VSCs) levels, organoleptic assessment of oral odor and the tongue-coating index were compared at baseline, 1, 5 and 9 hours after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Saudi Arabia volunteers to be recruited from Albaha province of Saudi Arabia via an online invitation on the e-learning blog www.alqumber.wordpress.com
2. No antibiotic usage and no antiseptic mouth rinse use for the last 3 months and one week preceding the commencement of the study, respectively.
3. Must be dentate healthy Saudi males aged 17-65 years, who adhere to the ritual of fasting.
4. provided informed consent form.

Exclusion Criteria:

1. Receiving any professional periodontal treatments (prophylactic scaling, root planning, and periodontal surgery) or professional advice during the previous year. 2. Prior to the inception of the study.

Ages: 17 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
viable anaerobic and aerobic bacterial counts | one month
  Measuring bacterial numbers by culturing of saliva samples
assessment of oral odor | one month
  the mouth odor was assisted by smelling
volatile sulfur compounds (VSCs) levels | one month
  these compound measured in part per million